CLINICAL TRIAL: NCT06881849
Title: Duration of Urinary Catheterization Following Cesarean Deliveries Under Neuraxial Anesthesia: A Prospective Cohort Study
Brief Title: Duration of Urinary Catheterization Following Cesarean Deliveries Under Neuraxial Anesthesia
Acronym: DUCC
Status: Not yet recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Anthony Chau, Clinical Associate Professor, University of British Columbia
Other Study IDs: H24-03410
Record Dates: First submitted 2025-02-13; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Cesarean Delivery; Urinary Catheterization
Keywords: patient recovery; cesarean delivery; urinary catheterization; foley catheter; patient anxiety

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In cesarean deliveries, urinary catheters are often used to help empty the bladder while patients have limited mobility. These catheters typically stay in during early recovery because certain pain medications can make it hard for patients to urinate. Recently, the Society of Obstetric Anesthesia and Perinatology (SOAP) recommended removing catheters within 6-12 hours after delivery to aid recovery. However, at BC Women's Hospital, a review found that catheters stayed in for an average of 19 to 19.4 hours, even when patients were mobile.

Leaving catheters in too long can increase the risk of urinary tract infections (UTIs), pain, and urination issues, which can delay recovery and extend hospital stays. An internal review showed that factors like patient anxiety may affect when catheters are removed. Postpartum anxiety affects around 9.9% to 20.7% of new mothers in the first year and is an important factor in recovery after a cesarean delivery.

The main goal of this study is to look at how long urinary catheters stay in patients who had a cesarean delivery under spinal or epidural anesthesia, and what the score is from a questionnaire used to measure anxiety called the State Trait Anxiety Inventory (STAI-S), to see if there is a link between them.

DETAILED DESCRIPTION:
This study aims to analyze how long foley catheters stay in the patient after their cesarean delivery under neuraxial anesthesia and what barriers there are in taking them out earlier.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥19 years of age.
* Undergoing cesarean delivery (elective or emergent) at BC Women's Hospital.
* Neuraxial anesthesia as their primary mode of anesthesia (spinal, epidural, combined spinal-epidural, dural-puncture epidural).
* In-patient status at 24 (+/- 8) hours.
* Self-reported proficiency in speaking and reading English.

Exclusion Criteria:

* Refusal to participate.
* Inability to provide informed consent.
* Other surgery (i.e. cervical cerclage) or delivery modes (i.e. operative vaginal delivery).
* De novo general anesthetic, or patients who had a conversion from neuraxial to a general anesthetic.
* Communication from patient's nurse indicating that it is not appropriate to approach due to distressing birth experience and/or outcome.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient's who underwent a cesarean delivery at BC Women's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-04-25 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between duration of urinary catheterization and STAI-S score | From the time of enrollment until urinary catheter removal, assessed up to 24 (+/- 8) postpartum.
  The STAI-S scale measures the respondents current state of anxiety by using terms to evaluate subjective feelings of worry, apprehension, concern, and nervousness. The scoring is 20-37 to indicate low anxiety, 38-44 to indicate moderate anxiety, and 45-80 to indicate high anxiety.

SECONDARY OUTCOMES:
Timing of delivery | From urinary catheter placement until its removal, assessed up to 24 (+/- 8) hours postpartum, categorized based on delivery time (e.g., morning: 06:00-11:59, afternoon: 12:00-17:59, evening/night: 18:00-05:59)
  This outcome measures the duration of urinary catheterization in relation to the time of delivery. Specifically, it examines whether the time of day a patient delivers (e.g., morning vs. afternoon vs. evening/night) is associated with differences in the length of time the urinary catheter remains in place. The duration of catheterization will be recorded in hours from placement to removal and compared across delivery time categories
Neuraxial Technique | From urinary catheter placement until its removal, assessed up 24 (+/- 8) hours postpartum, categorized by neuraxial technique used during delivery
  This outcome measures the duration of urinary catheterization in relation to the neuraxial anesthesia technique used for delivery. Specifically, it examines whether different neuraxial techniques (e.g., spinal, epidural, combined spinal-epidural, or dural-puncture epidural) are associated with differences in the length of time the urinary catheter remains in place. The duration of catheterization will be recorded in hours from placement to removal and compared across neuraxial technique groups
Opioid Dose | From urinary catheter placement until its removal, assessed up to 24 (+/- 8) hours postpartum, categorized by total neuraxial opioid dose administered.
  This outcome measures the duration of urinary catheterization in relation to the total opioid dose administered during neuraxial anesthesia for delivery. Specifically, it examines whether higher or lower opioid doses are associated with differences in the length of time the urinary catheter remains in place. The duration of catheterization will be recorded in hours from placement to removal and analyzed in relation to the opioid dose received during cesarean delivery. These opioid doses will be taken down: Total dose of spinal bupivacaine (mg), total dose of spinal fentanyl (mcg), total dose of spinal morphine (mg), total dose of epidural lidocaine (mg), total dose of epidural fentanyl (mcg), total dose of epidural morphine (mg).
Nursing Perception | Survey completed by the patient's postpartum nurse within 24 (+/- 8) hours after urinary catheter removal.
  This outcome measures postpartum nurses' perceptions of barriers to early urinary catheter removal. Nurses will complete a brief survey assessing nine predefined factors that may contribute to delayed catheter removal. Specifically, 'patient had difficulty mobilizing and/or voiding', 'patient had pain', 'patient was fatigued', 'patient experienced emotional and/or psychological distress', 'patient went to the NICU', 'patient requested to keep catheter in', 'patient had a history of infection (such as UTIs)', 'patient had a history of urinary retention', and 'concern about patient requiring re-catheterization'. Responses will be recorded as "Yes" or "No" for each statement, and the overall distribution of responses will be analyzed to identify common perceived barriers.

CONTACTS AND LOCATIONS:
Overall Officials: Anton Chau, MD MMSc, Principal Investigator — University of British Columbia
Locations (1):
- BC Women's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Figueiredo B, Conde A. Anxiety and depression in women and men from early pregnancy to 3-months postpartum. Arch Womens Ment Health. 2011 Jun;14(3):247-55. doi: 10.1007/s00737-011-0217-3. Epub 2011 Apr 9. PMID 21479759
- [Background] Julian LJ. Measures of anxiety: State-Trait Anxiety Inventory (STAI), Beck Anxiety Inventory (BAI), and Hospital Anxiety and Depression Scale-Anxiety (HADS-A). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11(0 11):S467-72. doi: 10.1002/acr.20561. No abstract available. PMID 22588767
- [Background] Goodman JH, Watson GR, Stubbs B. Anxiety disorders in postpartum women: A systematic review and meta-analysis. J Affect Disord. 2016 Oct;203:292-331. doi: 10.1016/j.jad.2016.05.033. Epub 2016 Jun 1. PMID 27317922
- [Background] Sutherland E, Yang T, Chau A. Duration of Urinary Catheterization After Cesarean Deliveries: A Retrospective Cohort Study..Poster session presented at: 2023 Summer Student Poster Day; 2023 Jul 27; Chieng Family Atrium, BC Children's Research Institute
- [Background] Bollag L, Lim G, Sultan P, Habib AS, Landau R, Zakowski M, Tiouririne M, Bhambhani S, Carvalho B. Society for Obstetric Anesthesia and Perinatology: Consensus Statement and Recommendations for Enhanced Recovery After Cesarean. Anesth Analg. 2021 May 1;132(5):1362-1377. doi: 10.1213/ANE.0000000000005257. PMID 33177330
- [Background] Basbug A, Yuksel A, Ellibes Kaya A. Early versus delayed removal of indwelling catheters in patients after elective cesarean section: a prospective randomized trial. J Matern Fetal Neonatal Med. 2020 Jan;33(1):68-72. doi: 10.1080/14767058.2018.1487394. Epub 2018 Jul 18. PMID 29886771

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2025-02-05): https://cdn.clinicaltrials.gov/large-docs/49/NCT06881849/Prot_SAP_000.pdf
  • Informed Consent Form: Patient Informed Consent Form (2025-02-05): https://cdn.clinicaltrials.gov/large-docs/49/NCT06881849/ICF_001.pdf
  • Informed Consent Form: Nurse Informed Consent Form (2025-02-05): https://cdn.clinicaltrials.gov/large-docs/49/NCT06881849/ICF_002.pdf